CLINICAL TRIAL: NCT05166551
Title: The Effect of Acupressure on Interventional Pain in Infancy Period Before Immunization: A Randomized Placebo-Controlled Trial
Brief Title: Effect of Acupressure on Interventional Pain in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tanju OĞUL, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Effect of Acupressure on Pain
Record Dates: First submitted 2021-12-14; First posted 2021-12-22 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Procedural Pain; Child, Only
Keywords: Infant; Procedural Pain; Acupressure
MeSH Terms: conditions — Pain, Procedural | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Acupressure will be applied to the infants in this group by the researcher in accordance with the technique for 1 minute on the GB31 acupuncture point on the leg where the vaccine will be administered.The considerations before, during and after acupressure application are as follows:
  * The hands will be washed to warm them up to body temperature.
  * The acupressure will be applied using the thumb to the GB31 acupuncture point for 1 minute before the vaccine is administered to the infants in the experimental group.
  * Pain scoring will be performed using the FLACC scale by the parents, the observing nurse, and the researcher after the vaccination procedure. In addition, the HR and SPO2 level of the infants before, during and after the procedure will be evaluated and recorded by the researcher.The crying time of infants will also be recorded.
  Interventions: Procedure: Acupressure
- Placebo Group (Placebo Comparator): Pressure will be applied by the researcher on a placebo point at least 2 cun above the GB31 acupuncture point, on the leg to be vaccinated, for 1 minute. The considerations before, during and after pressure are as follows:
  * The hands will be washed to warm them up to body temperature.
  * For the infants in the placebo group, pressure will be applied using the thumb for 1 minute to a placebo point that does not coincide with any acupuncture point at least 2 cun above the acupuncture point before the vaccine is administered.
  * Pain scoring will be performed using the FLACC scale by the parents, the observing nurse, and the researcher after the vaccination procedure. In addition, the HR and SPO2 level of the infants before, during and after the procedure will be evaluated and recorded by the researcher.The crying time of infants will also be recorded.
  Interventions: Procedure: Placebo Acupressure
- Control Group (No Intervention): The considerations before, during and after are as follows:
  Without any intervention, the infants in this group pain scoring will be performed using the FLACC scale by the parents, the observing nurse, and the researcher after the vaccination procedure. In addition, the HR and SPO2 level of the infants before, during and after the procedure will be evaluated and recorded by the researcher.The crying time of infants will also be recorded.

INTERVENTIONS:
Procedure: Acupressure — This study will be conducted in a randomized placebo-controlled research design to investigate the effect of acupressure, to be applied to the Gall Bladder (GB) 31 "Fengshi" acupuncture point before the vaccinations, on interventional pain in infants (0-1 years) caused by the vaccine.
  Arms: Experimental Group
Procedure: Placebo Acupressure — Placebo Acupressure
  Arms: Placebo Group

SUMMARY:
This study will be conducted to investigate the effect of acupressure, to be applied to the GallBladder (GB) 31 "Fengshi" acupuncture point before the vaccinations, on interventional pain caused by the vaccinations in infants. Considering the literature, it can be seen that acupressure is used in many fields and it's among the non-pharmacological methods that have been used by nurses in recent years.However, no study has been found to be conducted on the effect of acupressure, applied before the vaccine, on interventional pain caused by the vaccinations in infants. Therefore, this study aims to investigate the effect of acupressure applied before the vaccination on interventional pain in infants.

DETAILED DESCRIPTION:
Aim: This study will be conducted in a randomized placebo-controlled research design to investigate the effect of acupressure, to be applied to the GB31 acupuncture point before the vaccinations, on interventional pain in infants (0-1 years) caused by the vaccine.

Introduction: As a non-pharmacological method originating from traditional Chinese medicine with a 5000-year history, acupressure is used in different parts of the world as a method of treatment (Gach, 1990, Pour, Ameri, Kazemi, & Jahani, 2017). There are some points in the body that have great potential for energy transmission and are known as acupuncture points. In acupressure therapy, the body's regulatory processes are stimulated by applying pressure using fingers to acupuncture points located on the surface of the skin. The same points are used in acupuncture and acupressure. While acupuncture is performed using a needle, acupressure is performed by hands to make gentle but firm pressure (Ahmedov, 2015, Gach, 1990, Özşar, 2006). Acupressure is a more acceptable form of therapy for pediatric age groups since it is a non-invasive procedure (Abbasoğlu et al., 2015). In addition, its low cost, lack of side-effects, and its nature not requiring specific abilities for application are also among the advantageous aspects of this therapy (Wang, Escalera, Lin, Maranets, & Kain, 2008).

This study will be conducted to investigate the effect of acupressure, to be applied to the GB31 acupuncture point before the vaccinations, on interventional pain caused by the vaccinations in infants. The GB31 acupuncture point is located on the lateral midline of the thigh, 7 cun [(depends on patient's height), in adults 1 cun = approximately 3.3 cm] above the transverse popliteal fold, the point where the tip of the middle finger comes into contact when the patient is standing and lying flat on his/her back and putting his/her hands on the sides.

Considering the literature, it can be seen that acupressure is used in many fields and it's among the non-pharmacological methods that have been used by nurses in recent years. In this context, according to some nursing studies of acupressure on children, acupressure was found to be effective in reducing nausea and vomiting in children with cancer (Jones, Isom, Kemper, & McLean, 2008, Yeh et al., 2012), relieving the side-effects of chemotherapy and reducing fatigue (Farideh Bastani, Khosravi, Borimnejad, & Arbabi, 2015), improving quality of sleep (Carotenuto, Gallai, Parisi, Roccella, & Esposito, 2013), relieving the symptoms of asthma (Liu & Chien, 2015), reducing physical stress (Das, Nayak, & Margaret, 2011), alleviating postoperative symptoms (Norheim, Liodden, & Howley, 2010), and alleviating interventional pain (Koç Özkan, Şimşek Küçükkelepçe, & Aydin Özkan, 2019, Oğul & Yilmaz Kurt, 2021, Pour et al., 2017). However, no study has been found to be conducted on the effect of acupressure, applied before the vaccine, on interventional pain caused by the vaccinations in infants. Therefore, this study aims to investigate the effect of acupressure applied before the vaccination on interventional pain in infants.

Study Population and Sampling: The study population consists of the infants (regardless of gender) followed for vaccination by the studied university hospital, under the routine immunization program of the Ministry of Health, and the study sample will consist of infants who meet the research inclusion criteria. A power analysis was performed in order to determine the sample size. In the study, the power analysis was performed using the Gpower v.3.1.9.4 program. The study conducted by Unesi, Sajed, & Sharifzadeh (2019) was used to calculate the sample size (Unesi, Sajed, & Sharifzadeh, 2019). In the study, the minimum number of samples required was found to be 35 in each group (Type I Error = .05, The Power of the Test= .90), with the expectation that there should be statistical significance between the FLACC pain scale points of the infants in the intervention and control groups during the procedure. The study was planned to be completed with a total of 105 infants, including 35 in the experimental group, 35 in the placebo group, and 35 in the control group.

Data Collection Method: The data will be collected by the researcher in the unit where the study is planned to be carried out.

The following will be used in the collection of data:

* Data Collection Form, prepared by the researcher to determine the demographic characteristics of the infant, the researcher was conducted in accordance with the literature (Abbasoglu et al., 2015, Ahmedov, 2015, Tugcu et al., 2015). Some of the informations for this form (such as week of gestation, gender and anthropometric measurements in birth) will be taken from the child's personal records.
* Face, Legs, Activity, Cry, Consolability (FLACC) scale to determine the pain score of the infant during the administration of the vaccine (after the vaccination),
* Pulse Oximeter Device for detecting oxygen saturation (SPO2) and heart rate (HR) before, during and after vaccination of infants,
* Weighing Instrument to determine the current weight of infants,
* Height Measuring Tape to determine the current height of infants,
* Head Circumference Measurement Tape to determine the current head circumference of infants,
* Stopwatch of a smartphone for determining the crying duration of infants

Experimental Group Data Collection: After measuring the height, weight, and head circumference of the infants in this group, which are fed before the procedure and allowed to calm down on their mother's lap, acupressure will be applied by the researcher on the GB31 acupuncture point, on the leg to be vaccinated, for 1 minute in accordance with the acupressure technique. Detailed descriptions of the acupressure application technique and how much pressure will be applied to the selected points will not be included in the study. The considerations before during and after acupressure application are as follows:

* Before the acupressure application, hands will be washed to warm them up to body temperature.
* In accordance with the literature, acupressure will be applied using the thumb to the GB31 acupuncture point (on the lateral midline of the thigh, 7 cun above the transverse popliteal fold, the point where the tip of the middle finger comes into contact when the patient is standing and lying flat on his back and putting his/her hands on the sides) for 1 minute before the vaccine is administered to the infants in the experimental group.
* Pain scoring will be performed using the FLACC scale by the parents, the observing nurse, and the researcher after the vaccination procedure. In addition, the HR and SPO2 level of the infants before, during and after the procedure will be evaluated and recorded by the researcher. Pulse oximeter will be used in the evaluation process.The crying time of infants will also be recorded. Stopwatch will be used in the evaluation process.
* In terms of the reliability of the research results, the vaccine administration will be carried out by the same nurse working in the vaccine unit.

Placebo Group Data Collection: After measuring the height, weight, and head circumference of the infants in this group, which are fed before the procedure and allowed to calm down on their mother's lap, pressure will be applied by the researcher on a placebo (sham) point at least 2 cun above the GB31 acupuncture point, on the leg to be vaccinated, for 1 minute.

The following are the considerations to be taken into account before, during, and after the pressure application:

* Before the acupressure application, hands will be washed to warm them up to body temperature.
* For the infants in the placebo group, pressure will be applied using the thumb for 1 minute to a point (sham point) that does not coincide with any acupuncture point at least 2 cun above the acupuncture point before the vaccine is administered.

After the infants in the placebo group are allowed to calm down on the mother's lap for 5 minutes, pain scoring will be performed using the FLACC scale by the parents, the observing nurse, and the researcher, after the vaccination procedure. In addition, the HR and SPO2 level of the infants before during and after the procedure will be evaluated and recorded by the researcher.Pulse oximeter will be used in the evaluation process.The crying time of infants will also be recorded.Stopwatch will be used in the evaluation process. In terms of the reliability of the research results, the vaccine administration will be carried out by the same nurse working in the vaccine unit.

Control Group Data Collection: The infants in this group will be fed before the procedure, their height, weight, and head circumference will be measured and they will be allowed to calm down on their mother's lap. Without any intervention, the infants in this group will be allowed to calm down on the mother's lap for 5 minutes, and pain scoring will be performed using the FLACC scale by the parents, the observing nurse, and the researcher, after the vaccination procedure. In addition, the HR and SPO2 level of the infants before, during and after the procedure will be evaluated and recorded by the researcher.Pulse oximeter will be used in the evaluation process.The crying time of infants will also be recorded.Stopwatch will be used in the evaluation process. In terms of the reliability of the research results, the vaccine administration will be carried out by the same nurse working in the vaccine unit.

ELIGIBILITY:
Inclusion Criterias:

* Being healthy
* To be older than 4 weeks
* To be less than 1 year old
* Parents' consent to participate in the study
* To be born between 38-42 gestational weeks
* To take part in the routine vaccination program of the Ministry of Health

Exclusion Criterias:

* Being a sick infant
* To be over 1 year old
* Have taken analgesics in the last 4 hours
* To be born lower than 37 gestational weeks
* Parents' don't consent to participate in the study

Ages: 5 Weeks to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Pain severity | Starting with the vaccination and up to 1 minute after the procedure
  The parents will informed about the FLACC pain scale and they will asked to mark the children's pain levels on the scale. In addition, the pain levels of the children will determined by the researcher and a nurse who is a specialist in pediatric nursing by using the same scale.

SECONDARY OUTCOMES:
Heart rate (HR) | Before (1 minute), during and after (1 minute) the procedure
  The heart rate of the infants will measured with hand portable pulse oximeter (Nellcor, Covidien, Made in USA) device before, during and after the procedure.
Peripheral oxygen saturation level (SPO2) | Before (1 minute), during and after (1 minute) the procedure
  The peripheral oxygen saturation levels of the infants will measured with hand portable pulse oximeter (Nellcor, Covidien, Made in USA) device before, during and after the procedure.
Criying time | After the procedure (1 minute)
  Children's crying time will measured using a smart phone (Apple, Iphone 6s plus, Assembled in China) stopwatch after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu GÖZEN, Ph.D, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Abbasoglu A, Cabioglu MT, Tugcu AU, Ince DA, Tekindal MA, Ecevit A, Tarcan A. Acupressure at BL60 and K3 Points Before Heel Lancing in Preterm Infants. Explore (NY). 2015 Sep-Oct;11(5):363-6. doi: 10.1016/j.explore.2015.07.005. Epub 2015 Jul 3. PMID 26242287
- [Background] Bastani F, Khosravi M, Borimnejad L, Arbabi N. The effect of acupressure on cancer-related fatigue among school-aged children with acute lymphoblastic leukemia. Iran J Nurs Midwifery Res. 2015 Sep-Oct;20(5):545-51. doi: 10.4103/1735-9066.164508. PMID 26457090
- [Background] Carotenuto M, Gallai B, Parisi L, Roccella M, Esposito M. Acupressure therapy for insomnia in adolescents: a polysomnographic study. Neuropsychiatr Dis Treat. 2013;9:157-62. doi: 10.2147/NDT.S41892. Epub 2013 Jan 24. PMID 23378768
- [Background] Das R, Nayak BS, Margaret B. Acupressure and physical stress among high school students. Holist Nurs Pract. 2011 Mar-Apr;25(2):97-104. doi: 10.1097/HNP.0b013e31820d784a. PMID 21325910
- [Background] Jones E, Isom S, Kemper KJ, McLean TW. Acupressure for chemotherapy-associated nausea and vomiting in children. J Soc Integr Oncol. 2008 Fall;6(4):141-5. PMID 19134445
- [Background] Koc Ozkan T, Simsek Kucukkelepce D, Aydin Ozkan S. The effects of acupressure and foot massage on pain during heel lancing in neonates: A randomized controlled trial. Complement Ther Med. 2019 Oct;46:103-108. doi: 10.1016/j.ctim.2019.08.004. Epub 2019 Aug 6. PMID 31519265
- [Background] Liu CF, Chien LW. Efficacy of acupuncture in children with asthma: a systematic review. Ital J Pediatr. 2015 Jul 7;41:48. doi: 10.1186/s13052-015-0155-1. PMID 26149519
- [Background] Norheim AJ, Liodden I, Howley M. Implementation of acupuncture and acupressure under surgical procedures in children: a pilot study. Acupunct Med. 2010 Jun;28(2):71-3. doi: 10.1136/aim.2009.002220. Epub 2010 May 10. PMID 20458123
- [Background] Tanju O, Fatma Yilmaz K. Effect of acupressure on procedural pain before heel lancing in neonates. J Tradit Chin Med. 2021 Apr;41(2):331-337. PMID 33825415
- [Background] Pour PS, Ameri GF, Kazemi M, Jahani Y. Comparison of Effects of Local Anesthesia and Two-Point Acupressure on the Severity of Venipuncture Pain Among Hospitalized 6-12-Year-Old Children. J Acupunct Meridian Stud. 2017 Jun;10(3):187-192. doi: 10.1016/j.jams.2017.04.001. Epub 2017 Apr 24. PMID 28712478
- [Background] Tugcu AU, Cabioglu T, Abbasoglu A, Ecevit A, Ince DA, Tarcan A. Evaluation of peripheral perfusion in term newborns before and after Yintang (EX-HN 3) massage. J Tradit Chin Med. 2015 Dec;35(6):642-5. doi: 10.1016/s0254-6272(15)30153-9. PMID 26742308
- [Background] Wang SM, Escalera S, Lin EC, Maranets I, Kain ZN. Extra-1 acupressure for children undergoing anesthesia. Anesth Analg. 2008 Sep;107(3):811-6. doi: 10.1213/ane.0b013e3181804441. PMID 18713889
- [Background] Yeh CH, Chien LC, Chiang YC, Lin SW, Huang CK, Ren D. Reduction in nausea and vomiting in children undergoing cancer chemotherapy by either appropriate or sham auricular acupuncture points with standard care. J Altern Complement Med. 2012 Apr;18(4):334-40. doi: 10.1089/acm.2011.0102. PMID 22515794
- [Background] Unesi Z , Sajed A, Sharifzadeh G R. The Effects of Manual Pressure on the Injection Site on Vaccination Pain Among Infants: A Two-Group Clinical Trial. Mod Care J. 2019;16(4):e95705. doi: 10.5812/modernc.95705.